CLINICAL TRIAL: NCT01761838
Title: The Underlying Mechanism of Spinal Manipulative Therapy and the Effect of Pain on Physical Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00027069
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Low Back Pain; Degeneration of Lumbosacral Intervertebral Disc; Muscle Weakness; Spine Stiffness
Keywords: spinal manipulative therapy; low back pain; experimental pain; spinal stiffness; lumbar multifidus; degeneration
MeSH Terms: conditions — Low Back Pain; Muscle Weakness | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SMT for low back pain patients (Experimental): To investigate the effects of high velocity, low amplitude lumbopelvic spinal manipulative therapy on spinal stiffness and back muscle activity.
  Interventions: Other: SMT for low back pain patients
- Asymptomatic arm (Other): To investigate the sequential changes in spinal stiffness and back muscle activity of asymptomatic participants over time without any intervention. Participants of this arm can volunteer for an additional experimental pain protocol after their third visit (at 1 week) to investigate the effects of experimental pain on the changes of spinal stiffness and back muscle activity using a randomized crossover design (injecting 5% hypertonic saline or 0.9% isotonic saline to the interspinous ligaments at L3 to L5 levels in random order in two additional visits).
  Interventions: Other: Pain induction (optional)
- Low back pain participants without SMT (Other): To investigate the temporal changes in lumbar disc diffusion within a 1-hour period without SMT
  Interventions: Other: Low back pain participants without SMT

INTERVENTIONS:
Other: SMT for low back pain patients — High velocity, low amplitude spinal manipulative therapy (HVLA-SMT) will be provided to the lumbopelvic region on both sides.
  Other Names: High velocity, low amplitude spinal manipulative therapy; spinal manipulation
  Arms: SMT for low back pain patients
Other: Pain induction (optional) — A randomized crossover design is used to investigate the changes in spinal stiffness and back muscle activity of asymptomatic participants following an experimental pain induction procedure. Specifically, asymptomatic participants attend two separate sessions 5 days apart. Participants will receive 0.3 ml of 5% hypertonic saline or 0.9% isotonic saline in random order into the interspinous ligaments at L3 to L5 levels. The resulting temporal changes in pain intensity, spinal stiffness and trunk muscle activity following saline injections will be monitored. During the second session, the participants will undergo the same procedures but with the previously unused saline concentration.
  Arms: Asymptomatic arm
Other: Low back pain participants without SMT — No treatment
  Arms: Low back pain participants without SMT

SUMMARY:
The purpose of this study is to compare changes in spinal stiffness and back muscle activity between spinal manipulative therapy (SMT) responders, non-responders and asymptomatic participants. Additionally, the investigators wanted to compare the amount of lumbar degeneration between SMT responders, non-responders and asymptomatic participants. This study also determines if the presence of pain modifies post-SMT spinal stiffness and back muscle activity.

DETAILED DESCRIPTION:
SMT is a common manual therapy for treating patients with mechanical low back pain (LBP). SMT is defined as a high velocity, low amplitude thrust technique. Specifically, the clinician stands beside a supine patient. The patient is passively side-bent towards the side to be manipulated. The clinician passively rotates the patient and then delivers a high velocity, low amplitude thrust to the anterior superior iliac spine in a posteroinferior direction. SMT is indicated for patients with LBP judged to have spinal hypomobility or malalignment. Recently, our collaborators have discovered that LBP subjects who benefit from SMT can be identified prior to treatment by a five-item clinical prediction rule. Compared to non-responders, those who respond to SMT have: 1) more than 30% decrease in the modified Oswestry Disability Index score, 2) a significant and immediate decrease in spinal stiffness, and 3) a concurrent change in lumbar multifidus muscle activity. Taken together, the physical changes experienced by SMT responders alone provide an unique opportunity to better understand the mechanisms underlying SMT.

Since spinal stiffness is an important physical indicator of SMT response, it is important to understand the causal relation between pain, paraspinal/trunk muscle activity and spinal stiffness. Although research has shown positive correlation between pain and muscle activity, and between paraspinal muscle activity and spinal stiffness, the causal relation between pain, paraspinal/trunk muscle activity and spinal stiffness remains unknown. Given this background, an induction of temporary benign experimental pain to asymptomatic individuals can help clarify such causal relation and improve our understanding of physical responses in responders following pain resolution by SMT.

ELIGIBILITY:
Inclusion Criteria:

* Self ambulatory participants with or without acute/chronic LBP. LBP is defined as pain or discomfort between costal margin and above the gluteal folds, with or without leg pain.
* All the included LBP participants must have modified Oswestry Disability Index score > 12%
* Have the ability to lie prone for at least 20 minutes.
* Asymptomatic participants should be free from LBP at the time of visit.

Exclusion Criteria:

* With medical 'red flag' conditions such as cancer, cauda equine syndrome, spinal infection, fracture or systemic disease
* History of arm surgery, shoulder or arm pain that may hinder the arm lifting in prone
* History of orthopedic or neurological surgery to the spine, pelvis or hips
* Inflammatory or active infective processes involving spine or shoulder
* Spondylolisthesis, ankylosing spondylitis, scoliosis of greater than 20 degrees (Cobb's angle)
* Pregnancy
* Osteoporosis
* Neurologic deficit or signs of nerve root compression
* Congenital spinal disorder (such as spina bifida),
* Participation in competitive sports more than 3 times per week
* History of spinal manipulation or lumbar multifidus stabilization exercise training within the past 4 weeks
* Additional exclusion criteria for asymptomatic participants include: back pain in the preceding year, or exceeding 1 week; missed at least 1 work day because of back pain; and consultation for a back problem.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change of Modified Oswestry Low Back Pain Disability Index | baseline, Day 3, and 1 week
  It is a questionnaire to assess the participants' perceived low back pain related functional disability.
Change of 11-point Numeric Pain Rating Scale | baseline, Day 3, and 1 week
  It is a scale to measure the perceived pain intensity by the participants.
Change in Body Pain diagram | Baseline, Day 3, and 1 week
  The diagram will be used to demarcate the location and area of symptoms

SECONDARY OUTCOMES:
Change in measurement of lumbar multifidus muscle thickness by rehabilitative ultrasound imaging | Baseline, Day 3, and 1 week
  Using the rehabilitative ultrasound imaging to measure lumbar multifidus muscle thickness at rest and during an automatic muscle contraction.
Change of spinal stiffness testing by a mechanical indentation machine | Baseline, Day 3, and 1 week
  The spinal stiffness of participants will be measured by a validated mechanical indentation machine. Briefly, a 60 N load will be applied to the third lumbar spinous process and the corresponding spinal tissue deformations will be measured. The spinal stiffness will be calculated from the force-displacement curve of each indentation.
Electromyography of trunk muscles | At the third visit (1 week from the baseline)
  Electromyography of abdominal and erector spinae muscles during spinal stiffness testing will be measured.
Magnetic resonance imaging of lumbar region for participants with low back pain | At the beginning and immediately after the first visit (an expected average of 1 hour apart)
  It records the anatomical features of the lumbar spine and the changes in lumbar disc diffusion during the first session (an expected average of 1-hour duration).
Fear Avoidance Beliefs Questionnaire | Baseline
  It assesses the fear avoidance behaviour of participants
Change in Borg Category-Ratio Scale of Perceived Exertion | Baseline, Day 3, and 1 week
  It measures the subjective perception of exertion during the spinal stiffness test and muscle testings
Global Rating Of Change | 1 week after baseline
  It measures the perceived change of body function from the first visit.

OTHER OUTCOMES:
Measurement of lumbar multifidus muscle thickness by rehabilitative ultrasound imaging in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  Using the rehabilitative ultrasound imaging to measure lumbar multifidus muscle thickness at rest and during an automatic muscle contraction.
Spinal stiffness assessment by mechanical indentation machine in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  The spinal stiffness of participants will be measured by a validated mechanical indentation machine. Briefly, a 60 N load will be applied to the third lumbar spinous process and the corresponding spinal tissue deformations will be measured. The spinal stiffness will be calculated from the force-displacement curve of each indentation.
Electromyography of trunk muscles in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  Electromyography of abdominal and erector spinae muscles during spinal stiffness testing will be measured.
11-point Numeric Pain Rating Scale in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  It is a scale to measure the perceived pain intensity by the participants.
Body Pain diagram in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  The diagram will be used to demarcate the location and area of symptoms
Modified Oswestry low back pain disability index in the pain induction experiment | Before the injection in each session
  It is a questionnaire to assess the participants' perceived low back pain related functional disability.
Fear of Pain Questionnaire - III in the pain induction experiment | Before the injection in the first session
  It measures the perceived fear of pain under different hypothetical painful experiences.
Fear Avoidance Beliefs Questionnaire in the pain induction experiment | Before the injection in the first session
  It assesses the fear avoidance behaviour of participants
Borg Category-Ratio Scale of Perceived Exertion in the pain induction experiment | Before the injection, immediately after the injection, and 25-minute after the injection in each session
  It measures the subjective perception of exertion during the spinal stiffness test and muscle testings

CONTACTS AND LOCATIONS:
Overall Officials: Gregory N Kawchuk, PhD, DC, Principal Investigator — Department of Physical Therapy, Faculty of Rehabilitation Medicine, University of Alberta
Locations (1):
- River Valley Health Clinic, Edmonton, Alberta, Canada